CLINICAL TRIAL: NCT02092246
Title: Accuracy of Ultrasound Guided Versus Unguided Intra-articular Knee Injections in a Difficult to Inject Population
Brief Title: Ultrasound Guided vs Unguided Intra-articular Knee Injections
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty enrolling subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew Pingree, Assistant Professor of Physical Medicine and Rehabilitation, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-008328
Record Dates: First submitted 2014-03-13; First posted 2014-03-20 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis; Inflammatory Arthritis
MeSH Terms: conditions — Osteoarthritis; Arthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound Machine Guided Injection (Active Comparator): Use of ultrasound machine guidance in needle placement into the knee joint
  Interventions: Device: Ultrasound machine
- Unguided Injection (Active Comparator): Needle placement performed without ultrasound machine guidance
  Interventions: Device: Unguided injection

INTERVENTIONS:
Device: Ultrasound machine — Use of ultrasound machine guidance for accurate needle placement into the knee joint
  Other Names: Philips CX-50 Ultrasound Machine; FUJUFILM SonoSite X-Porte Ultrasound Machine
  Arms: Ultrasound Machine Guided Injection
Device: Unguided injection — Needle placement will take place without ultrasound machine guidance
  Other Names: Philips CX-50 Ultrasound Machine; FUJIFILM SonoSite X-Porte Ultrasound Machine
  Arms: Unguided Injection

SUMMARY:
To determine the accuracy of unguided versus ultrasound (US) guided knee joint injections in obese patients with no clinically detectable effusion.

DETAILED DESCRIPTION:
Patients with BMI > 30 and no clinically detectable knee effusions, with clinical symptoms and radiographic evidence of knee osteoarthritis or inflammatory arthritis, who have been referred for an intraarticular knee injection with corticosteroid will be randomized to either receive ultrasound guidance or not receive ultrasound guidance for their injection. One group will use the ultrasound guidance to position the needle. The other group will use landmarks to position the needle. For both groups, once the proceduralist is comfortable with needle placement for the injection, contrast dye will be injected and fluoroscopy used, to determine if the needle placement is correct. If it is determined the needle placement is not correct, fluoroscopy will be used to reposition it. Once needle placement is determined to be acceptable, the injection will be given. Patient demographics will be collected, along with pain scores preprocedure and two weeks post-procedure.

Subjects are responsible for all clinical costs associated with the injection.

There is no remuneration offered for study participation.

ELIGIBILITY:
Inclusion Criteria

* BMI > 30
* No clinically detectable knee effusion
* Clinical or radiographic evidence of knee osteoarthritis or inflammatory arthritis
* Must be referred to the Pain Clinic for treatment

Exclusion Criteria

* History of surgery on the affected knee
* Evidence of untreated systemic infection or systemic immunocompromise
* Evidence of cutaneous infections near the study knee injection site
* Patients on warfarin with an INR > 3.0
* Patients on oral antiplatelet or anticoagulant medications will be excluded if they have documented evidence of renal insufficiency (GFR < 60)
* History of iodinated contrast allergy or significant reaction to corticosteroids or lidocaine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the initial needle placement into the knee joint. | During the initial needle placement, which can take 1-5 minutes
  The number of participants with accurate initial needle placement into the knee joint

SECONDARY OUTCOMES:
Improved clinical efficacy of US guided knee injections compared to unguided knee injections | 30 minutes post injection
  Comparison of VAS scores 30 minutes after injection between subjects who had ultrasound guided knee injections and those who didn't

OTHER OUTCOMES:
Detection of knee effusions | During procedure, which can take up to 30 minutes to complete
  Comparison of the accuracy of detecting a knee effusion on clinical examination versus ultrasonographically

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Pingree, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States